CLINICAL TRIAL: NCT06860191
Title: Evaluation of the Effects of Different Root Canal Sealer and Irrigation Agitation Methods on Postoperative Pain in the Treatment of Teeth with Chronic Apical Periodontitis - Prospective Randomized Clinical Trial
Brief Title: Effect of Different Sealers and Activation Methods on Pain
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ipek Eraslan Akyuz, Research assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/1
Record Dates: First submitted 2025-02-01; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Chronic Apical Periodontitis
Keywords: Caries; apical periodontitis; irrigation agitation; root canal sealer
MeSH Terms: conditions — Periapical Periodontitis | interventions — Root Canal Filling Materials

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ah plus+MDA (Experimental): Ah plus will be used as the root canal sealer and manual dynamic activation will be used for irrigation agitation.
  Interventions: Drug: Root Canal Sealants
- Ah plus+PUA (Experimental): Ah plus will be used as the root canal sealer and pasive ultrasonic agitation will be used for irrigation agitation.
  Interventions: Drug: Root Canal Sealants
- Neosealer Flo+MDA (Experimental): Neosealer Flo will be used as the root canal sealer and manual dynamic activation will be used for irrigation agitation.
  Interventions: Drug: Root Canal Sealants
- Neosealer Flo+PUA (Experimental): Neosealer Flo will be used as the root canal sealer and pasive ultrasonic agitation will be used for irrigation agitation.
  Interventions: Drug: Root Canal Sealants

INTERVENTIONS:
Drug: Root Canal Sealants — In this study, different irrigation agitation methods and different root canal sealers will be compared.

SUMMARY:
In this study, the effects of different irrigation agitation methods and different root canal filling sealers on postoperative pain after root canal treatment will be evaluated.

DETAILED DESCRIPTION:
Root canal obturation is fundamental to successful root canal treatment. The primary objectives of root filling are to inhibit the growth of residual microorganisms following chemomechanical disinfection, prevent apical and coronal microleakage, and facilitate periapical tissue healing through appropriate materials and techniques. However, the intricate anatomy of the root canal system, including dentinal tubules, irregularities, and accessory canals, presents significant challenges to attaining an ideal root filling. Typically, this procedure uses a combination of core materials, such as gutta-percha, and root canal sealer. Sealers fill the spaces between the core material and the canal walls, ensuring a comprehensive three-dimensional filling that isolates any remaining bacteria and mitigates the risk of recontamination, reducing the likelihood of apical periodontitis.

In addition to their sealing function, root canal sealers exhibit antimicrobial properties and biocompatibility, which vary depending on their chemical composition. They are categorized based on their components into bioceramic-based, calcium hydroxide-containing, glass-ionomer-based, resin-based, silicone-based, and zinc-oxide eugenol sealers. Among these, epoxy-resin-based sealers, such as AH Plus, are widely recognized for their favorable physical properties, including low solubility and dimensional stability, often serving as benchmark materials for the evaluation of alternative sealers. Although AH Plus, an epoxy-resin-based sealer, is widely used in root canal treatment, it can lead to inflammation and pain if it comes into contact with periodontal tissues. In contrast, today bioceramic-based root canal sealers are gaining popularity due to their advantageous bioactive properties. These include antibacterial activity facilitated by an alkaline pH, promoting apical healing through hydroxyapatite formation, dentine structure mineralization, and effective sealing capabilities. Due to their hydrophilic nature, fine particle size, and ability to promote mineralized tissue formation, calcium silicate sealers provide excellent adaptation to canal walls, ensuring an effective seal and contributing to the overall success of the treatment. NeoSealer Flo is a bioactive ceramic paste that is premixed and contains a fine grade of inorganic powder made from tricalcium and dicalcium silicate. It is radiopaque, free from resin, and non-discoloring, and was formulated to harden when moisture from dentinal tubules is present. It possesses antimicrobial properties in vitro due to its high initial pH.

Nickel-titanium systems are recognized for their safety and efficiency. However, no preparation system can eliminate gutta-percha and sealers from canal walls. To address this limitation, various techniques to more effectively remove residual materials from root canals. These systems aim to enhance canal disinfection, improve solution penetration into the apical delta and lateral canals, and mitigate resistant bacterial strains that complicate dentinal tubular disinfection. Manual dynamic agitation (MDA), passive ultrasonic agitation (PUA), and sonic agitation are among the most commonly utilized activation techniques. During root canal preparation, using gutta-percha matching the diameter of the final file creates a dynamic irrigation effect through hydrodynamic activity generated by its oscillation in the irrigation solution. The MDA technique enhances debridement by improving the interaction between the irrigant and canal walls. PUA, introduced as an activation technique in the final stage of root canal treatment, offers multiple advantages. Systems like Ultra X enhance debris removal, microorganism elimination, and smear layer cleaning through high-speed flow, allowing the irrigant to reach accessory canals effectively without causing dentin damage. PUA achieves this by transmitting acoustic energy via ultrasonic waves through an oscillating file or wire, inducing two key actions: acoustic streaming, which generates hydrodynamic forces, and cavitation, where vapor-filled bubbles form within the fluid. Combining PUA with irrigants such as NaOCl, EDTA, and CHX has proven highly effective against E. faecalis.

There is insufficient data on the efficacy of adding MDA or PUA to the final irrigation protocol on postoperative pain after the single-visit endodontic treatment in cases with chronic apical periodontitis. Furthermore, there is a study in the literature regarding the potential effects of calcium-silicate-based NeoSealer Flo on postoperative pain. The purpose of this study is to evaluate the effect of different irrigation agitation techniques used in conjunction with resin-based (Ah Plus) and calcium silicate-based (NeoSealer Flo) sealers on postoperative pain in the treatment of chronic apical periodontitis.

The first null hypothesis of this study is that there is no statistically significant difference in treatment success, pain intensity, or frequency of occurrence following single-visit root canal treatment using AH Plus and NeoSealer Flo. The second null hypothesis is that there will be no statistically significant difference in postoperative pain intensity between the irrigation agitation techniques (MDA and PUA).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years who are classified as medically healthy (ASA I or II),
* Teeth that do not need periodontal and prosthetic treatment, with a periapical index score between 2 and 4,
* Teeth with single root and canal diagnosed with asymptomatic apical periodontitis,
* Teeth that respond negatively to electric pulp test (Parkell) or cold test (Endo Ice; Coltene, Altstätten, İsviçre), without pain during percussion and palpation.

Exclusion Criteria:

* Teeth with PAI scores lower than 2
* Patients who had taken analgesics or anti-inflammatory drugs in the last 4 hours
* Diabetic, immunocompromised, pregnant or history of antibiotic use in the last month or patients receiving antibiotic prophylaxis
* Teeth with root resorption, immature, severe crown damage, calcified canals, and previous root canal fillings

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain symptoms of the patients will be evaluated with prepared questionnaires, and periapical lesion healing will be evaluated with periapical radiographs. A visual analog scale will be used to measure the degree of pain. | 1-4 months
  Performing clinical and radiographic follow-up and evaluation of the patient.A visual analog scale will be used to measure the degree of pain.

IPD SHARING:
Plan to Share IPD: No
It was decided that it was appropriate to keep participant information confidential until the study was completed.